CLINICAL TRIAL: NCT05086666
Title: A Phase 1b/2 Clinical Study to Evaluate the Safety and Tolerability of AZD4547 in Patients With Solid Tumors and Its Efficacy in Patients With Locally Advanced or Metastatic Urothelial Carcinoma With FGFR2/3 Gene Alterations
Brief Title: A Phase 1b/2 Clinical Study to Evaluate the Safety and Tolerability and Efficacy of AZD4547
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK091-201
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-06

CONDITIONS: Urothelial Carcinoma
Keywords: urothelial carcinoma; FGFR2/3
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — AZD4547

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urothelial Carcinoma with FGFR2/3 Gene Alterations (Experimental): Evaluate the Efficacy of AZD4547 in Urothelial Carcinoma Patients with FGFR2/3 Gene Alterations
  Interventions: Drug: AZD4547

INTERVENTIONS:
Drug: AZD4547 — In Phase 1b study, subjects will receive continuous twice daily dosing in 21-day cycles (no matter if missed doses or delays exist), with pre-set dose cohorts of 80 mg BID and 120 mg BID.
  In Phase 2, subjects will receive continuous twice daily dosing in 21-day cycles with the RP2D or other doses as determined by the investigator and sponsor.
  Other Names: ABSK091

SUMMARY:
Phase 1b clinical study to evaluate the PK of oral AZD4547 in Chinese patients and RP2D. Phase 2 study to evaluate the efficacy of AZD4547 in urothelial carcinoma patients with FGFR2/3 gene alterations.

DETAILED DESCRIPTION:
This study is an open-label, Phase 1b/2 clinical study. In the Phase 1b study, the safety and tolerability of AZD4547 in patients with advanced solid tumors will be evaluated, the PK of oral AZD4547 in Chinese patients and the recommended phase 2 dose (RP2D) will be determined, and the antitumor activity will be preliminarily assessed. In the Phase 2 study, the efficacy of AZD4547 at the recommended dose in patients with locally advanced or metastatic urothelial carcinoma with FGFR2/3 gene alterations (including mutations and/or fusions) will be evaluated, and the safety, tolerability, and PK of AZD4547 will be further evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 25, both male and female;
2. Patients with histologically confirmed, surgically unresectable locally advanced or metastatic uroepithelial carcinoma that may be accompanied by other histologic differentiation (<50% of the total, including adenoid, squamous, or more aggressive sarcomatoid/micropapillary differentiation)
3. ECOG PS (performance status) score of 0-2;
4. Expected survival of ≥ 3 months;
5. Acceptable organ functions satisfy the following laboratory test requirements, and the test results should be obtained within 14 d prior to the first dose for study treatment (no transfusion of blood or blood products within 14 d prior to the blood test and no correction with bone marrow hematopoietic stimulating factors):
6. Female or male subjects of childbearing potential must agree to take medically approved measures for contraception during and for 6 months after the end of the study treatment; female subjects of childbearing potential must have a negative blood β-HCG test within 7 d prior to first dosing and must be non-lactating;
7. Subjects must voluntarily participate in this clinical trial, understand the study procedures and be able to sign an informed consent form in writing.

Exclusion Criteria:

1. Known to be allergic to AZD4547 tablets or constituents;
2. Subjects have previously received selective FGFR inhibitors (in the case of multi-target inhibitors including FGFR, it is required to discuss with the sponsor to decide whether they can be included);
3. There have been other malignancies requiring treatment in the past 2 years (except for cured skin cancer, cervical carcinoma in situ, basal cell carcinoma, focal prostate cancer with a Gleason score of 6, and focal prostate cancer at low risk of recurrence with a Gleason score of 3+4 and treated for more than 6 months at screening);
4. There are unstable (those who clinically/radiologically stable for at least 4 weeks prior to signing the ICF and requiring no long-term corticosteroid treatment may be enrolled) or symptomatic CNS metastases (other than pia mater metastases), or pia mater metastases of any condition;
5. The investigator determines that there are significant factors influencing oral drug absorption, such as inability to swallow complete pills, any type of uncontrollable nausea and vomiting, residual stomach dysfunction after total gastrectomy or subtotal gastrectomy, short bowel syndrome after small bowel resection, active diarrhea or irritable bowel syndrome requiring medical attention;
6. Time to the end of prior other antineoplastic therapy from the time of receiving the first dose of the study drug: < 4 weeks for major surgical operations (allowing palliative treatment for localized lesions), radiation therapy (> 30% bone marrow exposure), conventional chemotherapy, targeted therapy, immunotherapy, other interventional clinical study therapy (< 6 weeks for treatment with nitrosoureas or mitomycin); < 2 weeks or 5 drug half-lives (whichever is shorter) for endocrine therapy, herbal or Chinese medicinal preparations with antitumor indications, or herbal or Chinese medicinal preparations with adjuvant antitumor therapeutic effects;
7. Patients not recovered to ≤ CTCAE Grade 1 from reversible adverse events due to prior antineoplastic therapy (except for toxicities of no clinical significance such as alopecia, skin hypopigmentation, etc.);
8. There is a persistent increase in serum phosphorus levels (> ULN) requiring treatment control within 14 d prior to the first dose for study treatment;
9. Patients are using, or have used, within 14 d prior to the first dose of study treatment, the following drugs/foods: CYP3A4, 2D6 strong inhibitors or inducers (including grapefruit juice, grapefruit hybrids, pomegranate, star fruit, pomelo, Seville oranges and juice or other processed products);
10. There are uncontrolled cardiovascular diseases or a history thereof
11. Patients are taking medications during screening that may cause prolonged QTc interval or torsades de pointes (see section 5.4.3). Patients should discontinue such drugs for at least 5 d or 5 half-lives of the drug (whichever is longer) prior to the first dose for study treatment;
12. There are severe untreated skin/mucosal ulcers, chronic ulcers of the lower extremities, known gastric ulcers or incisions;
13. There is human immunodeficiency virus (HIV) infection (positive serologic test for HIV antibodies); active hepatitis B virus (HBV)/hepatitis C virus (HCV) infection (excluding those with a previous history of hepatitis C but a negative PCR test for hepatitis C virus during the screening period, or those with only positive hepatitis B virus surface antibodies on the hepatitis B test, or positive hepatitis B virus surface antigen but HBV DNA <1000 IU/mL);
14. There are any abnormal corneal or retinal changes during screening that may increase the risk of ocular toxicity
15. Any other medical (e.g., respiratory, metabolic, infectious, immune, congenital, endocrine, or central nervous system disorders), psychiatric, or social factors that may affect the subject's rights, safety, or the subject's ability to sign the informed consent form, cooperate, participate in the clinical study, or affect the interpretation of the study results as determined by the investigator.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-08-14 (Estimated); Study Completion 2024-05-27 (Estimated)

PRIMARY OUTCOMES:
DLT | 21 days
  Incidence of dose limiting toxicity (DLT)
AEs and SAEs | at least 6 months
  Incidence and grade of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI) (based on Common Terminology Criteria for Adverse Events, CTCAE 5.0) .
ORR | 6 months
  To confirm objective response rate (assessed by RECIST 1.1) in FGFR2/3 gene altered (including mutations and/or fusions) subjects with locally advanced or metastatic urothelial cancer with treated with AZD4547

SECONDARY OUTCOMES:
DOR | at least 6 months
  Duration of response (DoR): The time from the first evaluation of [CR] or [PR] until disease progression;
DCR | at least 6 months
  Disease control rate (DCR): DCR = [CR] + [PR] + stable disease [SD];
PFS | at least 6 months
  Progression-free survival (PFS): time to progression or death from the first day subjects receive AZD4547;

CONTACTS AND LOCATIONS:
Overall Officials: yuan lu, PhD, Study Director — Abbisko Therapeutics Co, Ltd
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China